CLINICAL TRIAL: NCT00950417
Title: Phase I Study of Nimotuzumab in Combination With Simultaneous Chemotherapy and Radiation for Patients With Locally Advanced Esophageal Cancer
Brief Title: Nimotuzumab in Combination With Chemoradiation for Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-ESO-T-0901
Record Dates: First submitted 2009-07-16; First posted 2009-07-31 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2009-07

CONDITIONS: Advanced Esophageal
Keywords: nimotuzumab esophageal chemo-radiotherapy
MeSH Terms: interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Esophageal Cancer (Experimental)
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab

SUMMARY:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The phase I study assessed the safety, and efficacy of the combination of Nimotuzumab administered concomitantly with chemo-radiotherapy in patients with locally advanced esophageal cancer tumours.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed before performing any of the study's specific procedures.
* ECOG performance status 0-2.
* Age > 18 and < 75.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, greater than or equal to 1 cm (longest diameter) by spiral computed tomography (CT) scan and MRI or greater than or equal to 2 cm by other ordinary radiographic technique.
* Histologically confirmed diagnosis of locally advanced esophageal.
* Life expectancy of more than 3 months.
* Use of an effective contraceptive method for patients of both sexes when there is a risk of conception and/or pregnancy.
* No serious blood producing,abnormal function of heart,lung, liver, or kidney or immuno-deficiency
* Neutrophils ≥3×109/L, platelet count≥100×109/L and haemoglobin≥9g/dL ,Creatinine ≤ 1.5 x NUL

Exclusion Criteria:

* Previous radiotherapy or chemotherapy
* Pregnant or breast-feeding women
* Drug abuse, unhealthy drug/alcohol addiction,or virus (HIV) infection
* Evidence of distant metastasis
* Participation in other clinical trials
* Patients with aphthosis, complete obstruction, fistula or deep peptic ulcer in the esophagus, or haematemesis
* Uncontrolled psychiatric disease or seizure
* Patients not fit for the clinical trial judged by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and toxicity of this new treatment. Both acute and chronic toxicity will be evaluated. | within study period

SECONDARY OUTCOMES:
To determine the complete response rate、partial rate、disease responserate、disease control rate in the patients subject to treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Chun Hu, Principal Investigator — Fu Dan University Cancer Hospital; Guo-Liang Jiang, Study Chair — Fu Dan University Cancer Hospital
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China